CLINICAL TRIAL: NCT02632643
Title: Assessment of the Efficacy of a Sensorimotor Approach After Maximum Three Sessions in Subjects With Symptomatic Temporomandibular Dysfunction (TMD) With Hypertonia: A Prospective, Multicenter Case Study.
Brief Title: Assessment of the Efficacy of a Sensorimotor Approach After Maximum Three Sessions in Subjects With TMD With Hypertonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Osteovox (Other)
Responsible Party: Principal Investigator, L'HOMME Sébastien, Dentist, Osteovox
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B707201525923
Record Dates: First submitted 2015-12-06; First posted 2015-12-17 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Temporomandibular Disorder
Keywords: TMD; HYPERTONIA; PARAFUNCTIONS; SENSORIMOTOR APPROACH
MeSH Terms: conditions — Temporomandibular Joint Disorders; Muscle Hypertonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counseling (Experimental)
  Interventions: Behavioral: Sensorimotor education with a view to obtaining an optimal FWS further to the relaxation of the masticatory, lingual and labial system. Learning of mandibular micro-movements in 5 directions.

INTERVENTIONS:
Behavioral: Sensorimotor education with a view to obtaining an optimal FWS further to the relaxation of the masticatory, lingual and labial system. Learning of mandibular micro-movements in 5 directions.

SUMMARY:
The study aims to demonstrate the efficacy of the sensorimotor approach developed by A. Piron (taught to the patient in three sessions) regarding three parameters related to TMD: facial pain, functional incapacities and hypertonia.

The subjects in the study are 18 to 77 years old and present the following conditions: a TMD disorder caused or aggravated by hypertonia and responsible for cervico-maxillo-facial pain and/or a functional incapacity in the last 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 77 years old.

Subjects presenting the following 3 characteristics:

1. A TMD disorder (objectivized by the DC/TMD 2014);
2. Facial pain in the last 30 days (objectivized by the Graded Chronic Pain Scale version 2.0 (GCPS v2.0)) and/or functional incapacity (chewing, mobility, verbal and emotional communication) in the last 30 days (objectivized by the Jaw Functional Limitation Scale 20 (JFLS-20));
3. Hypertonia (objectivized by the Oral Behaviors Checklist (OBC) short version and the Explanatory Model Scale).

Subjects who agree to comply with the requirements of the study. Subjects who are of age (and know how to read and write) who have given their informed, explicit consent in advance to any procedure related to the trial, the study or the investigation conducted on human beings, with the objective of developing knowledge specific to the exercise of health care professions, as set out in Royal Decree No. 78 of 10 November 1967 on the practice of the health care professions (Act of 27 December 2005).

Subjects insured under social security.

Exclusion Criteria:

* Any subject presenting at least one of the following criteria may not be included:
* Significant medical problems involving the following conditions:

Severe or progressive pathology (psychiatric, neurological, cardiopulmonary, renal, hepatic, endocrinological, hematological, neoplastic, infectious, metabolic or allergic).

Any acute trauma of the temporomandibular joint (trauma within the last 72 hours).

Severe anxiety or severe depression, as defined by a score greater than or equal to 15 on the HAD.

* Pregnant women
* Criteria related to prior or concurrent treatments:

Treatment with antipsychotics, anxiolytics, soporifics or muscle relaxants started within the two months preceding the study.

Treatment with intraoral implants during the study or in the two months preceding the study.

- Criteria related to lifestyle: Excessive alcohol consumption (WHO definition: more than two glasses per day for a woman and more than three for a man).

Subjects undergoing withdrawal or taking a replacement substance.

- Criteria related to the subject: Subjects unlikely, in the investigator's view, to comply with the instructions in the protocol.

Subjects unlikely, on the basis of a score <2 to question "C" of the Explanatory Model Scale, to comply with the therapy.

Subjects who had participated in a clinical trial in the previous month or were participating at the time of selection.

Subjects without the linguistic or psychological capacity to understand and sign the informed consent form and complete the psychometric questionnaires and psychological tests.

Exclusion criteria after acceptance in the study:

In addition to becoming aware a posteriori of an error related to the inclusion or exclusion criteria defined above, the therapist may decide to remove a subject before completion of the study.

The motivations for early exit are as follows:

* Subject who no longer agrees to comply with the requirements of the study.
* Occurrence of a major life stressor (score greater than 40 on the Holmes and Rahe Stress Scale).
* Need to redirect the subject to a different treatment. Any early exit from the study, whether decided on by the subject, the therapist or both together, will be recorded on a specific document, indicating the date and the reasons for the early exit.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall relief (from 0% to 100%) based on the ratio of "complaint after treatment" to "complaint before treatment". Multiple measurements related to both pain and functional incapacity are aggregated to arrive at one reported value: complaint | Beginning (day 0); during treatment (day 30 and day 90); end (day 180)
  Patient's complaint is calculated:
  * By integrating the weighting of both pain (P) and functional incapacity (FI) parameters in the complaint. 11 possibilities: [100% P - 0% FI] OR [90% P - 10% FI] OR [80% P - 20% FI] etc.
  * Patient's complaint = Pain and/or functional incapacity
  * Assessement of pain integrates 2 or 3 or 4 parameters: 2 are constant (intensity and frequency), 2 are optional (quality of life and drugs) because some painful patient don't take drug or don't have an altered quality of life. If there are 2 parameters, each = 50%; if 3 parameters, each = 33,3%; if 4 parameters, each = 25%
  * The scoring of the 4 pain parameters is based on questionnaires: Intensity: GCPS v2.0 (part 1): Score 0 to 100; Frequency (last month): Score 0 to 30; Drug: number of gram of the most specific medication (last month); Quality of life: GCPS v2.0 (part 2): score 0 to 6
  * Assessement of functional incapacity integrates 1 parameter: the JFLS-20 questionnaire (score from 0 to 200)

SECONDARY OUTCOMES:
Evidence of a change from baseline in the "intensity" component of cervico-maxillo-facial pain (a component of the primary outcome measure), on the basis of a questionnaire called "the Graded Chronic Pain Scale Version 2 (GCPS v2.0) (part 1)". | Beginning (day 0); during treatment (day 30 and day 90); end (day 180)
  3 Visual Analogic Scales (VAS) > 0 to 10. The scoring = the mean (0 to 100).
Evidence of a change from baseline in the "impact on quality of life" component of facial pain (a component of the primary outcome measure), on the basis of questionnaire called "the Graded Chronic Pain Scale Version 2 (GCPS v2.0) (part 2)". | Beginning (day 0); during treatment (day 30 and day 90); end (day 180)
  3 Visual Analogic Scales (VAS) > 0 to 10 and a 4th question about "how many days did pain keep the patient from doing usual activities" > 0 to 30 days.
  These 4 questions lead to a incapacity score from 0 to 6
Evidence of a change from baseline in the "frequency" component of facial pain (a component of the primary outcome measure), on the basis of a questionnaire developed by the authors. | Beginning (day 0); during treatment (day 30 and day 90); end (day 180)
  One question: "During the last 30 days, how many days did you have facial pain?" > 0 to 30 days
Evidence of a change from baseline in the "taking the most specific medication for painful attacks" component of facial pain (a component of the primary outcome measure), on the basis of a questionnaire developed by the authors. | Beginning (day 0); during treatment (day 30 and day 90); end (day 180)
  One question: "During the last 30 days, which drugs did you take to improve your facial pain?". Only one drug is taken into account: the most specific one used for facial pain > number of gram for the last month.
Evidence of a change from baseline in functional incapacity (a component of the primary outcome measure), on the basis of a questionnaire called " the Jaw Functional Limitation Scale (JFLS-20)". | Beginning (day 0); during treatment (day 30 and day 90); end (day 180)
  20 Visual Analogic Scales (VAS) > 0 to 10. The scoring = the sum (0 to 200).
Evidence of a change from baseline in oral behaviors induced by hypertonia, on the basis of a questionnaire developed by the authors and called "the short version of the Oral Behavior Checklist (OBC)". | Beginning (day 0); during treatment (day 30 and day 90); end (day 180)
  10 Visual Analogic Scales (VAS) > 0 to 4. The scoring = the sum (0 to 40).
Evidence of a change from baseline in dysacusis and feelings of dizziness, on the basis of a specific questionnaire developed by the authors. | Beginning (day 0) and end (day 180)
  7 Visual Analogic Scales (VAS) > 0 to 4. The scoring = the sum (0 to 28).
Evidence of a change from baseline in the patient's compliance with the treatment, on the basis of a questionnaire developed by the authors. | During treatment (day 30 and day 90) and end (day 180)
  2 Visual Analogic Scales (VAS) about both "observation" and "exercices" > 0 to 10.
  The scoring = the sum (0 to 20).
Evidence of the patient's subjective impressions of the treatment, on the basis of a questionnaire developed by the authors. | end (day 180)
  3 Visual Analogic Scales (VAS) about "difficulty of the treatment", "impact of the treatment on the long term" and "treatment easy to use in case of recurrence > 0 to 10.
  The scoring = the sum (0 to 30).
Evidence of correlations between the patient's psychological state (assessed with the HAD and SCL-90R) and the therapeutic efficacy of the approach (assessed by the patient's overall relief). | Beginning (day 0)
  2 questionnaires:
  * Hospital Anxiety and Depression Scale (HADS): 7 questions about anxiety (0 to 3)
    > Scoring = sum (0 to 21) and 7 questions about depression (0 to 3) > Scoring = sum (0 to 21).
  * Symptom Check-List (SCL 90 R): 90 questions about personality (0 to 4) > Scoring = 9 dimensions of the personality.
  See if there is a correlation between psychological state and therapeutic efficacy
Evidence of correlations between the patient's psychological state (assessed with the HAD and SCL-90R) and compliance with the treatment (assessed with a numerical scale created by the team in anticipation of the study). | Beginning (day 0)
  2 questionnaires:
  * Hospital Anxiety and Depression Scale (HADS): 7 questions about anxiety (0 to 3)
    > Scoring = sum (0 to 21) and 7 questions about depression (0 to 3) > Scoring = sum (0 to 21).
  * Symptom Check-List (SCL 90 R): 90 questions about personality (0 to 4) > Scoring = 9 dimensions of the personality.
  See if there is a correlation between psychological state and compliance
Evidence of the percentage of subjects diagnosed as hypertonic among all the patients diagnosed as having TMD (whether or not included in the study) by tracking the patients with a flowchart developed by the authors. | end (day 180)
  flowchart filled in by all investigators. At the top of the flowchart: all patients diagnosed TMD. The flowchart integrates all hypertonic patients. See the ratio: hypertonic TMD patients / All TMD patients.

CONTACTS AND LOCATIONS:
Overall Officials: L'HOMME Sébastien, Dentist, Principal Investigator
Locations (6):
- Belgium (3):
  - Cabinet de Logopédie Liesens-Denis, Berneau, Liège
  - Cabinet d'Ostéopathie PIRON, Beyne-Heusay, Liège
  - Cabinet de groupe LHR, Saive, Liège
- Cabinet d'Ostéopathie Garcion, Nantes, Loire-Atlantique, France
- Italy (2):
  - ANTONIO BIANCO Ortodontista e Osteopata, Gussago Bs, Brescia
  - Osteopata MARCO SBARBARO, Robassomero, Torino